CLINICAL TRIAL: NCT00795795
Title: Randomized Controlled Trial (RCT) of Preimplantation Genetic Screening (PGS) in Women of Advanced Maternal Age (AMA)
Brief Title: Preimplantation Genetic Screening in Women of Advanced Maternal Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Dr Carmen Rubio, Instituto Valenciano de Infertilidad
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0802-C-046-CR
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Chromosomal Abnormalities
Keywords: Chromosomal abnormalities in preimplantation embryos
MeSH Terms: conditions — Chromosome Aberrations | interventions — Phosphatidylglycerols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- with PGS (Active Comparator): IVF cycles with Preimplantation Genetic Screening (PGS)
  Interventions: Procedure: Preimplantation Genetic Screening
- Without PGS (Active Comparator): IVF cycle without Preimplantation Genetic Screening
  Interventions: Procedure: Preimplantation Genetic Screening; Procedure: IVF without PGS

INTERVENTIONS:
Procedure: Preimplantation Genetic Screening — Preimplantation Genetic Screening
Procedure: IVF without PGS — IVF without PGS
  Arms: Without PGS

SUMMARY:
An increased incidence of aneuploid pregnancies has been reported in women of advanced maternal age, with higher miscarriage rates. Cytogenetic studies in preimplantation embryos have shown elevated aneuploidy rate, particularly in women over 38 years. For these reasons, PGS has been applied to these patients to improve ongoing implantation rates, and most importantly, to decrease the risk of further miscarriages and affected offspring. In the past two years, several RCT have raised the question whether PGS is benefitial or not in AMA patients.

In our experience, PGS outcome in these patients offers higher ongoing implantation rates than the previously published in RCT studies, where no benefits for PGS were found. In these papers, poor technical skills, as well as unclear patients selection could explain the reported lack of PGS benefits.

Therefore, the objective of the present RCT is to analyze the outcome of IVF cycles with and without PGS in two age groups:

* Patients 38-39 years of age: 200 cyles per arm reaching embryo transfer should be performed
* Patients 40-44 years of age: 120 cycles per arm reaching embryo transfer Sample size has been calculated according to our retrospective experience with higher differences in ongoing implantation rates between cycles with and without PGS in patients of 40-44 years of age. In all patients embryo transfer will be performed on day 5. In the PGS group one cell will be biopsy in embryos with ≥5 cells on day-3 and chromosomes 13, 15, 17, 18, 21, 22, X and Y will be analyzed in two rounds. In the third round, nuclei with undoubtful or non-conclusive results will be analyzed using subtelomeric probes.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients over 37 years old, attending a fertility clinic

Exclusion Criteria:

* Azoospermic partners
* Female patients with uterine malformations
* number of retreived oocytes below 5

Ages: 38 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ongoing implantation per embryo and per pacient | one month

SECONDARY OUTCOMES:
Take home baby | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Valencia, Spain